CLINICAL TRIAL: NCT05724615
Title: Default Bulk Ordering and Text Messaging to Enhance Outreach for Lipid Screening
Brief Title: Default Bulk Ordering and Text Messaging to Enhance Outreach for Lipid Screening (Missing Lipids)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 852867
Record Dates: First submitted 2023-01-30; First posted 2023-02-13 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Atherosclerotic Cardiovascular Disease
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Intervention Model Description: This is a multilevel, pragmatic, 3-arm randomized clinical trial to assess completion of lipid panel testing. We will identify primary care patients eligible for lipid screening and randomize them in a 1:2:2 ratio to one of three arms during the intervention phase testing approaches requiring different degrees of p patient and clinician effort:
  Arm 1: Usual care Arm 2: Outreach + Bulk ordering Arm 3: Outreach + Bulk ordering + Text Based Reminders and Scheduling assistance
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual care (No Intervention): Participants will receive usual care only, and no additional intervention from this study.
- Outreach + Bulk ordering (Experimental): Participants will receive a standard mailed letter about lipid panel screening signed by Penn Primary Care, similar to birthday letters that are currently sent to some practices. These letters or messages will describe the importance of getting a lipid panel, their eligibility for a lipid panel, and information about fasting implications of getting the test. This letter will be complemented by a lipid panel order on behalf of their primary care provider, with a signed laboratory slip/order for lipid panel screening. Laboratory orders will be generated through bulk ordering in the electronic health records for all patients by a designated practice representative and the primary care provider as the authorizing clinician. Participants in Arm 2 will be asked to take the laboratory order to the laboratory of their choice to complete their test within the next 6 weeks.
  Interventions: Behavioral: Outreach + Bulk ordering
- Outreach + Bulk ordering + Text Based Reminders and Scheduling assistance (Experimental): Participants will receive a standard mailed letter, a signed laboratory slip/order, and text-based outreach. It will provide the patient information on walk-in hours in a partnering lab / or ask the patient to schedule an appointment with one of the listed Penn Labs with instructions on how to do so. Patients with an active MyPennMedicine account will be asked to schedule an appointment via MPM. Other patients will be sent a list with the contact of nearby available labs and opening hours and asked to call to schedule an appointment. Up to 2 reminder text messages with the deadline for the lab order will be sent to patients for which no appointment has been scheduled on MyPennMedicine at 2 weeks intervals. Enrollment in the text messaging platform will be opt-out. All results for lipid panel testing will be routed to the patients' primary care provider
  Interventions: Behavioral: Outreach + Bulk ordering + Text Based Reminders and Scheduling assistance

INTERVENTIONS:
Behavioral: Outreach + Bulk ordering — Participants will be sent an order for their lab screening and the recourse of the labs where they can schedule the screening.
  Arms: Outreach + Bulk ordering
Behavioral: Outreach + Bulk ordering + Text Based Reminders and Scheduling assistance — Participants will be sent an order for their lab screening and the recourse of the labs where they can schedule the screening. They will also receive text messages to remind them to have their lab completed as well as a link to schedule the lab and inform them of walk-in hours.
  Arms: Outreach + Bulk ordering + Text Based Reminders and Scheduling assistance

SUMMARY:
We aim to evaluate different approaches to increase Lipid screenings among primary care patients at Penn Medicine. A randomized trial will test the effectiveness of bulk ordering, outreach via mailed letters, and text-based reminders with scheduling assistance for patients needing a lipids panel. We will observe the number of completed panels after 3 and 6 months.

DETAILED DESCRIPTION:
Atherosclerotic cardiovascular disease (ASCVD) is a leading cause of mortality and disability in the United States. In order to prevent, predict and reduce ASCVD risk, clinicians will frequently use pool cohort equations (10 years CVD risk) to risk stratify patients and address modifiable risk factors. The American College of Cardiology/American Heart Association recommends routinely assessing traditional cardiovascular risk factors and calculation of 10-year ASCVD risk for adults 40 to 75 years of age and assessing traditional ASCVD risk factors for all adults 20 to 39 years of age at least every 4-6 years (Arnett et al., 2019 ). Among the components involved in the ASCVD risk stratification tool is a comprehensive lipid panel.

A mini-pilot on 100 patients overdue for lipid screening showed that bulk-ordering and text message concierge service (reminders and answering questions/concerns) increased response rate (21%) compared to conventional outreach (12%) or bulk-ordering only (9%). Qualitative analysis suggested that bulk-ordering as a default option reduces patient and clinician effort, and that uptake can benefit from trust enhancement (PCP endorsement), salience of communication (time-limited components, physical lab order), and effort/cognitive load reduction (text message reminders, scheduling assistance).

The aim is to conduct a pragmatic trial to evaluate the effect of bulk orders and text-based reminders on lipid screening rates among eligible patients who are overdue.H1: We hypothesize that reducing effort required from patients and clinicians through bulk ordering as a default with a reminder will result in greater completion of lipid screening compared to usual care.H2: We hypothesize that reducing effort through bulk ordering and providing complementary communication modalities (text message reminders and scheduling assistance) will result in higher response rates compared to bulk order and usual care.The primary study endpoint is the completion of the lipid panel within 3 months. An additional endpoint includes the number of patients with an elevated ASCVD risk score and the number of patients that had a clinical change (i.e. statin prescription) due to this information. The primary hypotheses are that Outreach + Bulk ordering (arm 2) will increase completion of lipid panel compared to usual care (arm 1), and that Outreach + Bulk ordering + Text Based Reminders (arm 3) will increase completion of lipid panel compared to usual care (arm 1) or conventional outreach + bulk ordering (arm 2). The results of the trial will also provide data that can be used to design future interventions that test the use of various behavioral economics tools to incentivize completion of lab tests. Secondary outcomes include completion of the lipid panel within 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are overdue for a lipid panel according to Health Maintenance in the EHR record (no lipid panel in the past 5 years or e those with diabetes or an annual lipid check modifier without a lipid panel for more than 1 year).
* Has PCP listed and at least 1 visit in last 3 years

Exclusion Criteria:

* Patients who do not have a cell phone listed in the EHR.
* Patients who have medical conditions that would significantly reduce likely benefit from lipid screening (metastatic cancer, hospice, palliative care).
* Preferred lab outside of Penn

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2023-12-07 (Actual)

PRIMARY OUTCOMES:
Number of participants that completed a lipid panel | 3 months from initial outreach
  Completion of lipid panel within 3 months across the 3 study arms.

SECONDARY OUTCOMES:
Number of participants that completed a lipid panel in the follow up period | 6 months from initial outreach
  Completion of lipid panel within 6 months across the 3 study arms.
AVCSD risk score | 6 months
  Proportion of patients with ASCVD risk score <5%(low risk), 5-7.5%(borderline risk), >=7.5%-<20% (intermediate risk) >=20%(high risk)
Patients initiated on statins | 6 months
  Proportion of patients initiated on statins once score is calculated

CONTACTS AND LOCATIONS:
Overall Officials: Shivan Mehta, MD, MBA, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pollak C, Parambath A, Coratti S, Norton L, Girard A, Reitz C, Snider CK, Xu L, Walker Z, John A, Putt ME, Volpp KG, Mehta SJ. Default Bulk Ordering and Text Messaging to Enhance Outreach for Lipid Screening: A Randomized Clinical Trial. JAMA Cardiol. 2025 Apr 1;10(4):313-320. doi: 10.1001/jamacardio.2024.5281. PMID 39879069